CLINICAL TRIAL: NCT02212808
Title: A Multicenter, 3-Stage Cluster Randomized Historically-Controlled Crossover Trial to Determine the Feasibility and Outcomes From Two Antimicrobial Stewardship Interventions in Community Hospitals
Brief Title: Antimicrobial Stewardship in Community Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052362; 1UM1AI104681-01 (NIH)
Record Dates: First submitted 2014-08-01; First posted 2014-08-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Antibiotic Stewardship in Community Hospitals
Keywords: Cluster-randomized crossover trial; Antimicrobial stewardship; Community hospitals; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antimicrobial restriction (Experimental): All prescriptions for targeted antibiotics will require phone approval by the trained PharmD during this arm. Prescribers will be instructed to contact the pharmacist via pager or phone call to discuss the patient details and the rationale for the desired antimicrobial. The pharmacist will then decide if the targeted antibiotic is approved or denied. If the pharmacist denies the use of the targeted antibiotic, the pharmacist will provide recommendations for alternative antibiotics for the specific clinical scenario.
  Interventions: Other: Antimicrobial restriction
- Post-antimicrobial prescription review (Experimental): All prescriptions for targeted antibiotics will be reviewed by the study pharmacist approximately 72 hours after initially written. The pharmacists will review a list of patients receiving the targeted antibiotics on a daily basis to identify patients who have received one or more targeted antibiotics for 72 hours (± 24 hours). The pharmacist will review and document the patient's current symptoms, pertinent clinical data, and the indication for the targeted antibiotic documented in the chart. Based on this review, the pharmacist will decide if the targeted antibiotic is necessary and/or if it needs to be modified. If a change is recommended, the pharmacist will then contact the prescriber to discuss the pharmacist's recommendations.
  Interventions: Other: Post-antimicrobial prescription review

INTERVENTIONS:
Other: Antimicrobial restriction — All prescriptions for targeted antibiotics will require phone approval by the trained PharmD during this arm. Prescribers will be instructed to contact the pharmacist via pager or phone call to discuss the patient details and the rationale for the desired antimicrobial. The pharmacist will then decide if the targeted antibiotic is approved or denied. If the pharmacist denies the use of the targeted antibiotic, the pharmacist will provide recommendations for alternative antibiotics for the specific clinical scenario. The pharmacist will document this interaction in the REDCap database.
  Arms: Antimicrobial restriction
Other: Post-antimicrobial prescription review — All prescriptions for targeted antibiotics will be reviewed by the study pharmacist approximately 72 hours after initially written. The pharmacist will review and document the patient's current symptoms, pertinent clinical data, and the indication for the targeted antibiotic documented in the chart. Based on this review, the pharmacist will decide if the targeted antibiotic is necessary and/or if it needs to be modified. If a change is recommended, the pharmacist will then contact the prescriber to discuss the pharmacist's recommendations. The interaction will be documented in the REDCap database.
  Arms: Post-antimicrobial prescription review

SUMMARY:
The Infectious Diseases Society of America (IDSA) guidelines recommend two "core" strategies for Antibiotic Stewardship (AS): 1) antimicrobial restriction and preauthorization and 2) prospective audit with intervention and feedback. Community hospitals have limited or no resources and staff dedicated to AS. Thus, understanding which of the core strategies is most feasible and effective in this practice setting would assist in appropriate allocation of limited resources. The purpose of this study is to evaluate the feasibility of implementing antimicrobial restriction and preauthorization vs. post antibiotic prescription review in resource-limited community hospitals.

DETAILED DESCRIPTION:
This study is a three-stage cluster randomized historically controlled crossover trial designed to evaluate the feasibility of the implementation of two AS strategies. Four community hospitals in the Duke Infection Control Outreach Network (DICON) will be recruited for this study. Ideally, hospitals will have no teaching affiliation, bed size <300, and no existing antimicrobial formulary restriction and preauthorization or post-antibiotic prescription review practices in place at study start.

Data will be obtained from the four community hospitals in three stages. In stage 1, historical data from each hospital will be collected for the year prior to study initiation from all participating hospitals. These data are used as a control representing current practice. In stage 2, the four hospitals will be divided into two pairs based upon bed size. One hospital from each pair will be randomly assigned to a six-month period of antimicrobial restriction and preauthorization (Strategy 1; stage 2) followed by a six-month period of post-antibiotic prescription review (Strategy 2; stage 3). The other two hospitals will undergo Strategy 2 in stage 2 followed by Strategy 1 in stage 3 to help alleviate the concern for seasonal/temporal effects when comparing the strategies to each other. A one-month wash out will be performed between each stage. Three antibiotics will be specifically targeted for intervention: anti-pseudomonal carbapenem of choice at the study hospital, vancomycin, and piperacillin-tazobactam. Utilization of alternative antimicrobials, including fluoroquinolones, cephalosporins, and anti-methicillin resistant Staphylococcus aureus (anti MRSA) systemic antimicrobials (e.g., nafcillin, daptomycin, linezolid, ceftaroline, clindamycin, and trimethoprim-sulfamethoxazole (TMP-SMX)) will also be collected. All study hospitals will have electronic systems that track antimicrobial prescriptions through orders, electronic medication administration records (eMAR), bar-coded medication administration (BCMA), or dispensing data.

Hospitals will have dedicated clinical pharmacist time for preauthorization or post-antibiotic review for the three targeted antibiotics in each arm of the study. Pharmacists (PharmDs) at each site will receive standardized training by study personnel in order to address common questions and anticipated arguments, and to establish a robust knowledge base regarding the targeted antimicrobials (anti-pseudomonal carbapenem of choice at the study hospital, vancomycin, and piperacillin-tazobactam). They will also be trained in conflict management.

Study personnel will provide suggested criteria for appropriate use of each targeted drug. Hospital P&T committees will review, edit (if desired), and approve hospital-specific protocols for appropriate use criteria for each study drug. Pharmacists will be provided with specific clinical pathways for urinary tract infections (UTIs), community-acquired pneumonia (CAP), healthcare-associated pneumonia (HCAP), bacteremia, and "other" uses of targeted antimicrobial. Clinical pathways will be developed jointly by study personnel and based on Centers for Disease Control and Prevention pilot projects. Clinical pharmacists will determine appropriateness of therapy based on study clinical pathways, their baseline knowledge, and acquired knowledge derived by training from study personnel. Time spent performing the two stewardship strategies will be supported by grant funds. The designated pharmacist will be involved in two critical components of the protocol: a) completing the intervention and b) documenting the outcome of the intervention.

ELIGIBILITY:
Inclusion Criteria:

-All adult and pediatric patients admitted to the study hospital who are prescribed targeted or alternative antimicrobial agent(s) will have data collected from their medical records.

Exclusion Criteria:

* Any patient not meeting the criteria above will be excluded.
* Patients who receive < 24 hours of surgical prophylaxis with a targeted or alternative antimicrobial will be excluded.
* Finally, any patient followed by an Infectious Disease consultant will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3972 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility 1 - Intervention Approval | Prior to implementation, estimated length of 3 months up to 6 months
  To evaluate administrative steps required for protocol approval of two stewardship intervention strategies at study hospitals.
Feasibility 2 - PharmD training | Prior to implementation, estimated length of 1 months up to 2 months
  To evaluate the steps required for training of local PharmD(s) to administer the two stewardship strategies.
Feasibility 3 - PharmD Time | Day of Intervention, expected length of 20 hours per week up to 52 weeks
  To estimate and compare the time required of the pharmacist to administer the different strategies.
Feasibility 4 - Resource Utilization | During hospitalization, an expected length of 14 days, up to 30 days
  To estimate and compare the resource utilization of each strategy, including pharmacist time and cost of antibiotics.

SECONDARY OUTCOMES:
Antimicrobial utilization - Days of Therapy | During Hospitalization, an expected length of 14 days, up to 30 days
  To compare the total days of therapy of targeted and alternative antibiotics between each strategy.
Patient Outcomes | During Hospitalization, an expected length of 14 days, up to 30 days
  To compare patient-specific outcomes between each strategy including but not limited to total hospital days, death and ICU admission
Pharmacist/Physician Perceptions | Within 1 month of completion of intervention arm
  To compare the prescriber and pharmacist perceptions of the two stewardship strategies

CONTACTS AND LOCATIONS:
Overall Officials: Deverick J Anderson, MD, MPH, Principal Investigator — Duke University

REFERENCES:
- [Derived] Anderson DJ, Watson S, Moehring RW, Komarow L, Finnemeyer M, Arias RM, Huvane J, Bova Hill C, Deckard N, Sexton DJ; Antibacterial Resistance Leadership Group (ARLG). Feasibility of Core Antimicrobial Stewardship Interventions in Community Hospitals. JAMA Netw Open. 2019 Aug 2;2(8):e199369. doi: 10.1001/jamanetworkopen.2019.9369. PMID 31418804